CLINICAL TRIAL: NCT02302846
Title: Phase II Study Of Ixazomib As Maintenance Therapy For Patients With Acute Myeloid Leukemia (AML) And High Risk Myelodysplastic Syndrome (MDS) In Remission
Brief Title: Study of MLN9708 as Maintenance Therapy for Patients With Acute Myeloid Leukemia (AML) and High Risk Myelodysplastic Syndrome (MDS) in Remission
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Millennium: The Takeda Oncology Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0379; NCI-2014-02604 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2014-11-18; First posted 2014-11-27 (Estimated); Results first posted 2018-10-03 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Leukemia
Keywords: Leukemia; Acute myeloid leukemia; AML; High-risk myelodysplastic syndrome; MDS; Ixazomib; MLN9708
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute | interventions — ixazomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ixazomib (Experimental): Participants receive 4 mg oral dose of Ixazomib on Days 1, 8 and 15 of each 28-day cycle.
  Interventions: Drug: Ixazomib

INTERVENTIONS:
Drug: Ixazomib — 4 mg by mouth on Days 1, 8 and 15 of each 28-day cycle.
  Other Names: MLN9708

SUMMARY:
The goal of this clinical research study is to learn if ixazomib can prevent AML or MDS from coming back in patients who are in remission. The safety of this drug will also be studied.

DETAILED DESCRIPTION:
Study Drug Administration:

Each study cycle is 28 days.

If you are found to be eligible to take part in this study, you will take ixazomib capsules on Days 1, 8 and 15 of each cycle. Ixazomib capsules should be swallowed whole, with water, on an empty stomach (take the dose at least 1 hour before or 2 hours after a meal).

If you miss a dose, take it as soon as you remember, as long as the next scheduled dose is more than 3 days away. If you vomit after taking a dose, do not make up the dose but continue with the next scheduled dose as planned.

You may receive the study drug for up to 12 cycles. If the doctor thinks it is in your best interest, you may be able to continue taking the study drug beyond Cycle 12.

Study Visits:

On Day 1 of each cycle (+/- 1 day):

* You will have a physical exam.
* Blood (about 2-3 teaspoons) will be drawn for routine tests.

On Days 8 and 15 of Cycle 1, blood (about 2-3 teaspoons) will be drawn for routine tests.

Every third cycle, you will have a bone marrow aspiration and/or biopsy to check the status of the disease.

Length of Study:

You may continue taking the study drug for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over after the end-of-study visit.

End-of-Study Visit:

After your last dose of study drug, you will return to the clinic for an end-of-study visit.

* Blood (about 2-3 tablespoons) will be drawn for routine tests.
* You will have a bone marrow aspirate and/or biopsy to check the status of the disease.

This is an investigational study. Ixazomib is not FDA-approved or commercially available. It is currently being used for research purposes only. The study doctor can explain how the study drug is designed to work.

Up to 40 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 18 years of age or older.
2. Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
3. Female patients who: Are postmenopausal for at least 1 year, OR Are surgically sterile, OR If they are of childbearing potential, agree to practice 2 effective methods of contraception, from the time of signing the informed consent through 90 days after the last dose of study drug, OR Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.) Male patients, even if surgically sterilized, must agree to one of the following: Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, OR agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject.
4. Patients must have a history of de novo or therapy-related AML (defined by World Health Organization (WHO) classification of >/= 20% bone marrow blasts) or high-risk MDS (defined by International Prostate Symptom Score (IPSS) or IPSS-R)
5. 5. Patients must be in a documented complete response/incomplete blood count recovery (CR/CRi) from either their front-line or first salvage therapy as evidenced by </= 5% bone marrow blasts and absence of extramedullary disease. (For patients with prior MDS who then transformed to AML, therapy received for MDS is not considered prior therapy for AML)
6. Patients should have received at least 2 cycles of induction therapy or 1 induction and 1 consolidation cycle, OR patient should be considered to have completed all planned chemotherapy, OR patient is considered to be unable, unfit or unwilling to receive additional chemotherapy.
7. Eastern Cooperative Oncology Group (ECOG) performance 0, 1, or 2.
8. Patients must meet the following clinical laboratory criteria: - Absolute neutrophil count (ANC) >/= 500/mm3 and platelet count >/= 50,000/mm3. Platelet transfusions to help patients meet eligibility criteria are not allowed within 3 days before study enrollment - Total bilirubin </= 1.5 x the upper limit of the normal range (ULN). - Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST)</= 3 x ULN. - Calculated creatinine clearance >/= 30 mL/min

Exclusion Criteria:

1. Female patients who are lactating or have a positive serum pregnancy test during the screening period.
2. Failure to have fully recovered (ie, </= Grade 1 toxicity) from the reversible effects of prior chemotherapy.
3. Major surgery within 14 days before enrollment.
4. Radiotherapy within 14 days before enrollment. If the involved field is small, 7 days will be considered a sufficient interval between treatment and administration of the MLN9708.
5. Known central nervous system involvement
6. Infection requiring systemic antibiotic therapy or other serious infection within 14 days before study enrollment.
7. Evidence of current uncontrolled cardiovascular conditions, including sustained hypertension (SBP >150mmHg on two or more readings one week apart without normalization in between), clinically significant uncontrolled cardiac arrhythmias, symptomatic Class III-IV New York Heart Association (NYHA) congestive heart failure, unstable angina, or myocardial infarction within the past 6 months.
8. Systemic treatment, within 7 days, or the half life of the treatment, whichever is longer before the first dose of MLN9708, with strong inhibitors of CYP1A2 (fluvoxamine, enoxacin, ciprofloxacin), strong inhibitors of cytochrome P CYP3A (clarithromycin, telithromycin, itraconazole, voriconazole, ketoconazole, nefazodone, posaconazole) or strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort.
9. Ongoing or active systemic infection, history of hepatitis B or C virus infection, or known human immunodeficiency virus (HIV) positive.
10. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
11. Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
12. Known GI disease or GI procedure that is expected to interfere with the oral absorption or tolerance of MLN9708 including difficulty swallowing. As determined by the investigator.
13. Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection
14. Patient has >/= Grade 3 peripheral neuropathy, or Grade 2 with pain on clinical examination during the screening period.
15. Administration of other investigational agents for the treatment of AML/MDS within 21days (or 5 times the terminal half life of the investigational treatment whichever is longer) of the start of this trial and throughout the duration of this trial.
16. At the time of registration, stem cell transplantation is not planned within the next 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-03-20 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Courtney DiNardo, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: May 2015 through March 2016. All participants recruited at The University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: Of the five participants enrolled in this study, three were evaluable for response. One participant was evaluable for toxicity. A fifty participant was registered but did not receive therapy due to the patient's decision to continue a prior therapy.
Period: Overall Study
Arm/Group | Ixazomib
Started | 5
Completed | 4
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ixazomib
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 2
Age, Continuous [Median (Full Range); unit: years] | 60 [20 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Relapse-Free Survival (RFS)
Description: RFS defined as interval from date of enrollment to date of first objective documentation of disease relapse or death from any cause. Survival or times to failure and time to progression functions estimated using Kaplan-Meier method.
Time Frame: 84 days
Population: Three participants were evaluable for response. One patient was evaluable for toxicity only. No other analysis is possible due to the low number of patients accrued.
Measure: Median (Full Range); unit: Weeks
Arm/Group | Ixazomib
Number analyzed (Participants) | 3
Weeks | 34 [19 to 50]

ADVERSE EVENTS:
Time Frame: Adverse events reported during each treatment course, an average of one year . Overall period: May 2015 to March 2016.
Arm/Group | Ixazomib
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ixazomib (N=4)
Fall (General disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ixazomib (N=4)
Intermittent Headache (General disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (3)
Dizziness (Nervous system disorders) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 1 (1)
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Decreased White Blood Count (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-11): https://cdn.clinicaltrials.gov/large-docs/46/NCT02302846/Prot_SAP_000.pdf